CLINICAL TRIAL: NCT06578299
Title: The Real World Study of First Line Treatment of HER2 Positive Recurrent/Metastatic Breast Cancer With Inetetamab Combined With Paclitaxel With/Without Pertuzumab（INTPOWER）
Brief Title: Inetetamab Combined With Paclitaxel With/Without Pertuzumab for Previously Treated HER2-positive Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Director of Phase I Clinical Trial Department; Professor, Chief physician of oncology department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTPOWER
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Inetetamab and Paclitaxel ± Pertuzumab Inetetamab：was administered as an intravenous (IV) loading dose of 8mg/kg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 6mg/kg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Paclitaxel：Docetaxel 75mg/m2, albumin paclitaxel 260mg/m2, or paclitaxel liposomes 175mg/m2) is administered intravenously on the first day of every three weeks, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Pertuzumab：was administered as an intravenous (IV) loading dose of 840mg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 420mg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inetetamab and Paclitaxel ± Pertuzumab (Experimental): Inetetamab and Paclitaxel ± Pertuzumab Inetetamab：was administered as an intravenous (IV) loading dose of 8mg/kg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 6mg/kg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Paclitaxel：Docetaxel 75mg/m2, albumin paclitaxel 260mg/m2, or paclitaxel liposomes 175mg/m2) is administered intravenously on the first day of every three weeks, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Pertuzumab：was administered as an intravenous (IV) loading dose of 840mg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 420mg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Interventions: Drug: Inetetamab and Paclitaxel ± Pertuzumab

INTERVENTIONS:
Drug: Inetetamab and Paclitaxel ± Pertuzumab — Inetetamab and Paclitaxel ± Pertuzumab Inetetamab：was administered as an intravenous (IV) loading dose of 8mg/kg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 6mg/kg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Paclitaxel：Docetaxel 75mg/m2, albumin paclitaxel 260mg/m2, or paclitaxel liposomes 175mg/m2) is administered intravenously on the first day of every three weeks, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Pertuzumab：was administered as an intravenous (IV) loading dose of 840mg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 420mg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.

SUMMARY:
This study is designed to comprehensively evaluate the HER2 positive recurrent/metastatic breast cancer patients in the real world who receive the combination of Inetetamab and Paclitaxel ± Pertuzumab, including basic characteristics, efficacy and safety. The results of this study are helpful to further understand the efficacy and safety of HER2 positive patients with recurrent/metastatic breast cancer who receive the combination of Inetetamab and Paclitaxel ± Pertuzumab in the first line, and help clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 70 years, female
2. Patients with HER2-positive breast cancer defined as immunohistochemical (IHC) test + + +, or FISH test positive
3. Participants must have histologically or cytologically confirmed invasive breast cancer with locally recurrent inoperable or radiological evidence of metastatic disease
4. Have not received first-line anti-HER2 treatment or (neo) adjuvant anti-HER2 drug treatment that is effective and has been discontinued for more than 12 months
5. Patients with assessable target lesion as per RECIST 1.1 and irRECIST criteria;
6. ECOG PS score 0 or 1, estimated survival time ≥3 months, and can be followed-up;
7. The cardiopulmonary function is basically normal, with LVEF ≥ 50%;
8. Adequate organ function;
9. Female patients of childbearing age who have negative pregnancy tests and voluntarily adopt effective and reliable contraceptive measures；
10. The patient voluntarily signs an informed consent form.

Exclusion Criteria:

1. Participated in other clinical trials within 4 weeks;
2. Have received any systematic anti-tumor treatment during the recurrence/metastasis stage (excluding endocrine therapy previously performed for recurrence/metastasis stage);
3. During the (neo) adjuvant phase, other anti-HER2 treatments were received in addition to trastuzumab and pertuzumab;
4. Patients who experience disease progression during (neo) adjuvant trastuzumab treatment, as well as patients who experience recurrence/metastasis within 12 months after completing (neo) adjuvant system treatment;
5. Evidence of central nervous system metastasis or leptomeningeal disease;
6. Individuals with a known history of allergies to the components of this medication regimen;
7. Pregnant or lactating women;
8. Left ventricular ejection fraction<50% for cardiac function; Patients with obvious clinical manifestations such as arrhythmia, myocardial ischemia, severe atrioventricular block, heart dysfunction, and severe heart valve disease;
9. The researchers believe that it is not appropriate to participate in this trial, as any other medical, social, or psychological factors may affect safety or compliance with research procedures.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
PFS | Until progression, assessed up to approximately 24 months
  PFS is defined as the time from the participant's first dose of study treatment to the first date of either disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Until progression, assessed up to approximately 24 months
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Clinical Benefit Rate (CBR) | Until progression or death, assessed up to approximately 24 months
  Clinical benefit rate was defined as the percentage of participants with confirmed best overall response of complete response (CR) or partial response (PR) or stable disease（SD）>6 months determined by investigator using RECIST v1.1 on two consecutive occasions ≥4 weeks apart.
Overall Survival (OS) | Up to approximately 3 years
  OS is defined as the time from the participant's first dose of study treatment to the date of death.
Number of Participants With Adverse Events (AEs) | Up to approximately 3 years
  Assessment of the toxicity profile of regimen according to the National Cancer Institute Common Toxicity Criteria version 5.0 (NCI CTCAE v 5.0).